CLINICAL TRIAL: NCT01466816
Title: Skeletal Muscle Lipid Metabolism and Insulin Sensitivity: Can Dietary Fatty Acid Composition Modulate Muscle Lipid Storage?
Brief Title: Lipids and Insulin Sensitivity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: 08-3-030
Record Dates: First submitted 2011-10-19; First posted 2011-11-08 (Estimated); Last update posted 2011-11-08 (Estimated); Status verified 2011-11

CONDITIONS: Obesity; Insulin Resistance
Keywords: Lipid metabolism
MeSH Terms: conditions — Obesity; Insulin Resistance

STUDY DESIGN:
Who Masked: Participant

ARMS (3):
- Saturated fatty acid test meal (Experimental)
  Interventions: Dietary Supplement: test meals with various fatty acid compositions
- Monounsaturated fatty acid meal (Experimental)
  Interventions: Dietary Supplement: test meals with various fatty acid compositions
- Polyunsaturated fatty acid meal (Experimental)
  Interventions: Dietary Supplement: test meals with various fatty acid compositions

INTERVENTIONS:
Dietary Supplement: test meals with various fatty acid compositions — Three different milkshakes with a U13C palmitate tracer added

SUMMARY:
Rationale: The investigators hypothesize that a change in dietary fat quality (an increase in unsaturated fatty acids) may modulate fuel partitioning within the type 2 diabetic muscle towards less accumulation of lipid metabolites and an improved insulin sensitivity.

Objective:

1. The contribution of dietary vs endogenous fat sources to lipid overflow in the circulation and to skeletal muscle lipid uptake and storage in obese insulin resistant subjects vs obese insulin sensitive controls.
2. The acute effect of meals with various fatty acid composition ((high saturated (SFA) vs polyunsaturated (PUFA) vs monounsaturated (MUFA)) on skeletal muscle lipid uptake and storage, fatty acid mediated gene expression and postprandial insulin sensitivity in obese insulin resistant subjects.

Study design: single-blind randomized cross-over trial

Study population: obese males (35-70 years) with or without insulin resistance

Intervention:

1. 1 test meal
2. 3 test meals with a different fatty acid composition

Main study parameters/endpoints:

More insight whether dietary fat quality may modulate circulating lipids and skeletal muscle fatty acids handling, and may affect oxidative capacity and lipid storage in parallel to an increased insulin sensitivity.

ELIGIBILITY:
Inclusion Criteria:

* Obese males aged between 35 and 70 years with insulin resistance.

Exclusion Criteria:

* History of type 2 diabetes.
* Liver or kidney failure.
* Diseases in which the live expectation is shorter then 5 years.
* The use of experimental medication.
* Diseases/medication use that may have an influence on the glucose tolerance.
* Not to be able to understand the study information.
* Users of fatty acid supplements including fish oils etc.
* Users of high doses of antioxidant vitamins.
* Athletes.
* People on a diet of people that are planning to lose weight.

Ages: 35 Years to 70 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2008-10; Primary Completion 2010-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Acute effect of meals with various fatty acid composition on postprandial insulin sensitivity | the individual participants will be measured within 8-10 weeks.
  The acute effect of meals with various fatty acid composition ((high saturated (SFA) vs polyunsaturated (PUFA) vs monounsaturated (MUFA)) on postprandial insulin sensitivity will be measured during the stable isotope test.
Acute effect of meals with various fatty acid composition on forearm muscle fatty acid handling | the individual participants will be measured within 8-10 weeks.
  Using the stable isotope technique, we can differentiate between the metabolic fate of dietary versus endogenous fatty acids

SECONDARY OUTCOMES:
Acute effect of meals with various fatty acid composition on intramuscular fatty acid handling | the individual participants will be measured within 8-10 weeks.
Acute effect of meals with various fatty acid composition on transcriptional regulation of the fatty acid metabolism in skeletal muscle biopsies | the individual participants will be measured within 8-10 weeks.
  Transcriptional regulation will be measured by means of microarray.

CONTACTS AND LOCATIONS:
Overall Officials: Ellen E Blaak, PhD, Prof, Principal Investigator — Maastricht University Medical Centre +
Locations (1):
- Maastricht University Medical Centre +, Maastricht, Limburg, Netherlands

REFERENCES:
- [Derived] Jans A, Konings E, Goossens GH, Bouwman FG, Moors CC, Boekschoten MV, Afman LA, Muller M, Mariman EC, Blaak EE. PUFAs acutely affect triacylglycerol-derived skeletal muscle fatty acid uptake and increase postprandial insulin sensitivity. Am J Clin Nutr. 2012 Apr;95(4):825-36. doi: 10.3945/ajcn.111.028787. Epub 2012 Feb 15. PMID 22338035